CLINICAL TRIAL: NCT02243982
Title: Predictive and Diagnostic Value of Tau and Beta-amyloid Markers in Cerebrospinal Fluid and Positron Emission Tomography in the Dementia of Parkinson's Disease
Brief Title: Predictive and Diagnostic Value of Tau and Beta-amyloid Markers in the Dementia of Parkinson's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Maria Jose Martí, MD, PhD, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI1080236
Record Dates: First submitted 2014-08-13; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2009-12

CONDITIONS: Parkinson's Disease; Parkinson-Dementia Syndrome
Keywords: Parkinson, dementia, FDDNP, tau, beta-amyloid
MeSH Terms: conditions — Parkinson Disease; Progressive supranuclear palsy atypical; Dementia; Pick Disease of the Brain; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [F18]-FDDNP (Experimental): 2-(1-{6-[(2-[fluorine-18]fluoroethyl)(methyl)amino]-2-naphthyl}-ethylidene)malononitrile. Radiopharmaceutical tracer
  Interventions: Other: [F18]-FDDNP

INTERVENTIONS:
Other: [F18]-FDDNP — radiopharmaceutical tracer, intravenous, single dose, of 360+/- 20 megabecquerel
  Other Names: 2-(1-{6-[(2-[fluorine-18]fluoroethyl)(methyl)amino]-2-naphthyl}-ethylidene)malononitrile

SUMMARY:
The PET tracer Fluoro-ethyl-methyl-amino-naphthyl-ethylidene-malononitrile ([F18]-FDDNP) has a specific affinity for lesions containing tau protein and beta-amyloid The study consists of two phases

* In a first transversal phase, 8 neurologically unimpaired controls, 15 patients with PD and no dementia (PDND) and 8 with PD and dementia (PDD) will undergo lumbar puncture for study of tau, phospho-tau and beta-amyloid levels in cerebrospinal fluid (CSF), as well as positron emission tomography (PET) with ([F18]-FDDNP. Concentration of CSF markers and both the degree and topography of FDDNP-PET uptake will be compared among groups, along with correlation analysis between CSF and PET findings.
* During the second phase (18 months follow-up), the PDND patients will undergo the same procedures, and cognitive changes including incident dementia will be assessed. The correlation between cognitive impairment and neurochemical and neuroimaging changes will be established to determine the predictive value of these markers.

Since the pathological lesions observed in Alzheimer disease (AD) are common in the PD and the concentrations of tau and beta-amyloid are altered in AD and PET with [F18]-FDDNP is able to separate patients with AD and cognitive impairment from controls, we hypothesized that:

1. - Patients with PD will show a biomarkers profile similar to the AD (decreased levels of beta-amyloid and increased phospho-tau and tau) in CSF, and an abnormal uptake of [F18]-FDDNP PET compared to PDND patients and controls.
2. -The distribution of cortical [F18]-FDDNP in the PD will be different from the AD and similar to dementia with Lewy bodies, predominantly in posterior cortical areas.
3. PDND patients will show a [F18]-FDDNP PET uptake and levels of protein markers in CSF intermediate between controls and patients with PD.
4. -In the subsequent follow-up, PDND patients will show cognitive impairment correlate to changes in the levels of protein markers in CSF and uptake of PET with [F18]-FDDNP
5. - The predictive value for the development of dementia in PD of specific patterns of PET uptake and CSF proteins profile will be established.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria PDD

* Male or female ≥ 60 years old;
* Diagnose of PD probable or definite according to criteria of the United Kingdom Parkinson's Disease Society Brain Bank;
* The Hoehn & Yahr stage of the disease between 3 and 5 in off state;
* Diagnose of dementia established according to the fourth edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and the diagnostic guidelines for dementia of the Movement Disorders Society (MDS);
* The score of the Mini-Mental State Examination of Folstein (MMSE) <24;
* The score on the Mattis Dementia Rating Scale (MDRS) <136.

Inclusion criteria PDND:

* Male or female ≥ 60 years old;
* Diagnose of PD probable or definite according to criteria of the United Kingdom Parkinson's Disease Society Brain Bank;
* The Hoehn & Yahr stage of the disease between 3 and 5 in OFF state;
* The score of the Mini-Mental State Examination of Folstein (MMSE) ≥24;
* The score on the Mattis Dementia Rating Scale (MDRS) ≥136.

Inclusion criteria Controls:

* Male or female ≥ 60 years old;
* No known diagnosis of neuropsychiatric diseases
* The score of the Mini-Mental State Examination of Folstein (MMSE) ≥24;
* The score on the Mattis Dementia Rating Scale (MDRS) ≥136.

Exclusion Criteria:

* The subject is pregnant or breastfeeding;
* The subject has a history of drug abuse or alcohol;
* The subject has developed dementia in the first year of parkinsonism or before than parkinsonism;
* The subject meets criteria for vascular dementia;
* The subject has symptoms suggestive of other types of parkinsonism (multi-system atrophy cortico-basal, supra-nuclear palsy progressive degeneration) or degenerative dementia (fronto-temporal dementia);
* The subject has a moderate or severe renal functional impairment (serum creatinine> 1.5 mg / dL);
* The subject has a moderate or severe hepatic impairment (bilirubin> 2 times the upper limit of normal, transaminases> 3 times the upper limit of normal);
* The subject presents structural abnormalities in basal ganglia or cortical level on magnetic resonance imaging or computerized tomography;
* The subject has participated in a clinical study with an investigational drug product within 30 days prior to screening and / or radiopharmaceutical in a minimum period of 5 radioactive half-lives prior to screening;
* Occupational exposure to radiation> 15 milliSievert (mSv) / year
* The subject has received treatment with non-steroidal anti-inflammatory drugs during the 30-day period before the PET scan
* The subject has allergy to the investigational product or any of its components;
* The subject has a clinically active, serious disease with a reduced life expectancy;
* The subject is claustrophobic / a.
* The subject has received in the last 364 days a dose of ionizing radiation that coupled with the study dose exceeds 10 mSv

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Relative Volume of Distribution of [F18]-FDDNP in non-demented patients with Parkinson's disease (PDND), demented patients with Parkinson's disease (PDD) and controls. | Baseline assessment
  To asses the [F18]-FDDNP PET uptake in non-demented patients with Parkinson's disease (PDND), demented patients with Parkinson's disease (PDD) and controls.

SECONDARY OUTCOMES:
Concentration ( pg/mL) of beta-amyloid, tau and phospho-tau in cerebrospinal fluid (CSF) of non-demented patients with Parkinson's disease (PDND), demented patients with Parkinson's disease (PDD) and controls. | Baseline assessment
  Enzyme linked immunosorbent assay (ELISA) method will be used to assess the concentration of the biomarkers in the CSF.
Number of patients without dementia at baseline that switch to dementia at 18 months follow-up | 18 months
  PDND group will be followed-up at 18 months to assess the number of patient that develops dementia, using the criteria of Diagnostic and Statistical Manual of Mental Disorders version IV.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose Martí, Md, PhD, Principal Investigator — Fundació per a la Recerca Biomedica
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Caballol N, Marti MJ, Tolosa E. Cognitive dysfunction and dementia in Parkinson disease. Mov Disord. 2007 Sep;22 Suppl 17:S358-66. doi: 10.1002/mds.21677. PMID 18175397
- [Background] Aarsland D, Perry R, Brown A, Larsen JP, Ballard C. Neuropathology of dementia in Parkinson's disease: a prospective, community-based study. Ann Neurol. 2005 Nov;58(5):773-6. doi: 10.1002/ana.20635. PMID 16240351
- [Background] Lashley T, Holton JL, Gray E, Kirkham K, O'Sullivan SS, Hilbig A, Wood NW, Lees AJ, Revesz T. Cortical alpha-synuclein load is associated with amyloid-beta plaque burden in a subset of Parkinson's disease patients. Acta Neuropathol. 2008 Apr;115(4):417-25. doi: 10.1007/s00401-007-0336-0. Epub 2008 Jan 8. PMID 18185940
- [Background] Jellinger KA, Wenning GK, Seppi K. Predictors of survival in dementia with lewy bodies and Parkinson dementia. Neurodegener Dis. 2007;4(6):428-30. doi: 10.1159/000107703. Epub 2007 Oct 9. PMID 17934326
- [Background] Blennow K, Hampel H. CSF markers for incipient Alzheimer's disease. Lancet Neurol. 2003 Oct;2(10):605-13. doi: 10.1016/s1474-4422(03)00530-1. PMID 14505582
- [Background] Jansen Steur E, Vermes I, de Vos RA. Cerebrospinal-fluid tau protein and aspartate aminotransferase in Parkinson's disease. Lancet. 1998 Apr 11;351(9109):1105-6. doi: 10.1016/s0140-6736(05)79387-9. No abstract available. PMID 9660591
- [Background] Mollenhauer B, Trenkwalder C, von Ahsen N, Bibl M, Steinacker P, Brechlin P, Schindehuette J, Poser S, Wiltfang J, Otto M. Beta-amlyoid 1-42 and tau-protein in cerebrospinal fluid of patients with Parkinson's disease dementia. Dement Geriatr Cogn Disord. 2006;22(3):200-8. doi: 10.1159/000094871. Epub 2006 Aug 7. PMID 16899997
- [Background] Fagan AM, Mintun MA, Mach RH, Lee SY, Dence CS, Shah AR, LaRossa GN, Spinner ML, Klunk WE, Mathis CA, DeKosky ST, Morris JC, Holtzman DM. Inverse relation between in vivo amyloid imaging load and cerebrospinal fluid Abeta42 in humans. Ann Neurol. 2006 Mar;59(3):512-9. doi: 10.1002/ana.20730. PMID 16372280
- [Background] Maetzler W, Reimold M, Liepelt I, Solbach C, Leyhe T, Schweitzer K, Eschweiler GW, Mittelbronn M, Gaenslen A, Uebele M, Reischl G, Gasser T, Machulla HJ, Bares R, Berg D. [11C]PIB binding in Parkinson's disease dementia. Neuroimage. 2008 Feb 1;39(3):1027-33. doi: 10.1016/j.neuroimage.2007.09.072. Epub 2007 Oct 22. PMID 18035558
- [Background] Agdeppa ED, Kepe V, Liu J, Flores-Torres S, Satyamurthy N, Petric A, Cole GM, Small GW, Huang SC, Barrio JR. Binding characteristics of radiofluorinated 6-dialkylamino-2-naphthylethylidene derivatives as positron emission tomography imaging probes for beta-amyloid plaques in Alzheimer's disease. J Neurosci. 2001 Dec 15;21(24):RC189. doi: 10.1523/JNEUROSCI.21-24-j0004.2001. PMID 11734604
- [Background] Shoghi-Jadid K, Small GW, Agdeppa ED, Kepe V, Ercoli LM, Siddarth P, Read S, Satyamurthy N, Petric A, Huang SC, Barrio JR. Localization of neurofibrillary tangles and beta-amyloid plaques in the brains of living patients with Alzheimer disease. Am J Geriatr Psychiatry. 2002 Jan-Feb;10(1):24-35. PMID 11790632
- [Background] Smid LM, Vovko TD, Popovic M, Petric A, Kepe V, Barrio JR, Vidmar G, Bresjanac M. The 2,6-disubstituted naphthalene derivative FDDNP labeling reliably predicts Congo red birefringence of protein deposits in brain sections of selected human neurodegenerative diseases. Brain Pathol. 2006 Apr;16(2):124-30. doi: 10.1111/j.1750-3639.2006.00006.x. PMID 16768752
- [Background] Small GW, Kepe V, Ercoli LM, Siddarth P, Bookheimer SY, Miller KJ, Lavretsky H, Burggren AC, Cole GM, Vinters HV, Thompson PM, Huang SC, Satyamurthy N, Phelps ME, Barrio JR. PET of brain amyloid and tau in mild cognitive impairment. N Engl J Med. 2006 Dec 21;355(25):2652-63. doi: 10.1056/NEJMoa054625. PMID 17182990
- [Background] Kepe V, Huang SC, Small GW, Satyamurthy N, Barrio JR. Visualizing pathology deposits in the living brain of patients with Alzheimer's disease. Methods Enzymol. 2006;412:144-60. doi: 10.1016/S0076-6879(06)12010-8. PMID 17046657
- [Background] Logan J, Fowler JS, Volkow ND, Wang GJ, Ding YS, Alexoff DL. Distribution volume ratios without blood sampling from graphical analysis of PET data. J Cereb Blood Flow Metab. 1996 Sep;16(5):834-40. doi: 10.1097/00004647-199609000-00008. PMID 8784228
- [Derived] Buongiorno M, Antonelli F, Compta Y, Fernandez Y, Pavia J, Lomena F, Rios J, Ramirez I, Garcia JR, Soler M, Camara A, Fernandez M, Basora M, Salazar F, Sanchez-Etayo G, Valldeoriola F, Barrio JR, Marti MJ. Cross-Sectional and Longitudinal Cognitive Correlates of FDDNP PET and CSF Amyloid-beta and Tau in Parkinson's Disease1. J Alzheimers Dis. 2017;55(3):1261-1272. doi: 10.3233/JAD-160698. PMID 27814297